CLINICAL TRIAL: NCT05794607
Title: Investigation of the Effectiveness of Tele-pulmonary Rehabilitation After Lung Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Halime Sinem Barutçu (Other Government)
Responsible Party: Sponsor-Investigator, Halime Sinem Barutçu, Physical Therapist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Organization: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DrLutfiKirdarPT
Record Dates: First submitted 2023-03-16; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Tele-pulmonary Rehabilitation; Lung Cancer; Lung Resection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who will undergo lung surgery for lung cancer
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Rehabilitation group
- Control group (No Intervention)

INTERVENTIONS:
Other: Rehabilitation group — The intervention group will be given strength training to improve muscle strength and flexibility, and aerobic exercise training to improve exercise capacity with function.
  Arms: Study group

SUMMARY:
As a result of the review in the literature, no study was found in which tele-pulmonary rehabilitation was applied after physiotherapist-supervised lung resection via video conferencing.

Therefore, in this study, it was planned to investigate the effectiveness of tele-pulmonary rehabilitation in patients diagnosed with lung cancer and undergoing lung resection.

DETAILED DESCRIPTION:
Research; It was planned as a prospective and randomized controlled study. The research universe is Istanbul Kartal Dr. Lütfi Kırdar City Hospital Chest Surgery Clinic will consist of cases with a preliminary diagnosis of lung cancer. The sample of the study, on the other hand, will consist of patients who agreed to participate in the study and who met the inclusion criteria, who were planned for lung resection.

1. Study group (n=18); The treatment features of the tele-pulmonary rehabilitation group via videoconferencing are; Within the scope of the tele-pulmonary rehabilitation program, an exercise program consisting of lower-upper extremity strengthening training and flexibility training, breathing exercises training (diaphragmatic breathing, thoracic expansion exercises and forced expiration) and aerobic exercise training will be created before discharge, exercise session will be followed. Re-evaluation will be done after 8 weeks.Exercise intensity will be planned as 2 days a week with supervision and 1 day without supervision, 3 days a week in total. Exercise safety will be ensured by taking the severity of shortness of breath of the patients as a reference.
2. Control group (n=18); Patients in the tele-pulmonary rehabilitation control group will be given respiratory and aerobic exercise advice before discharge. Re-evaluation will be done after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 55-75 years diagnosed with lung cancer
* Patients who underwent lobectomy, segmentectomy, bilobectomy, and pneumonectomy by either VATS or thoracotomy surgeries
* Patients who can use phones and make video calls

Exclusion Criteria:

* Patients with heart failure or atrial fibrillation
* Patients with acute infection at the time of assessment
* Patients who have had myocardial infarction in the last six months
* Patients with any comorbidities such as uncontrolled diabetes mellitus and/or hypertension
* Patients with any problem that would limit physical activity

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional exercises capacity | 8 weeks
  A 6-minute walk test will be performed to determine functional exercise capacity.
Pulmonary function test | 8 weeks
  Pulmonary function test will be made in accordance with ats criteria
Peripheral muscle strength | 8 weeks
  Peripheral muscle strength will be done with 'Lafayette' device
Upper extremity normal range of motion | 8 weeks
  Upper extremity normal range of motion will be measured with a manual goniometer

SECONDARY OUTCOMES:
Anxiety and depression | 8 weeks
  Hospital anxiety and depression scale (HAD scale); It will be used to measure and evaluate patients' anxiety and depression scales.
Determination of quality of life | 8 weeks
  EORTC QLQ-C30; This scale is a widely used quality of life scale in cancer patients all over the world.
Cognitive functions | 8 weeks
  Mini mental state test; will be used to evaluate postoperative cognitive dysfunction.

IPD SHARING:
Plan to Share IPD: Undecided